CLINICAL TRIAL: NCT01783821
Title: LIPS-B: Lung Injury Prevention Study With Budesonide and Beta Agonist (Formoterol)
Brief Title: LIPS-B: Lung Injury Prevention Study With Budesonide and Beta
Acronym: LIPS-B
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Stanford University (Other); Beth Israel Deaconess Medical Center (Other); University of Arizona (Other); National Center for Research Resources (NCRR) (NIH)
Responsible Party: Principal Investigator, Emir Festic, M.D., Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 12-008192; UL1RR024150 (NIH)
Record Dates: First submitted 2013-01-31; First posted 2013-02-05 (Estimated); Results first posted 2016-09-05 (Estimated); Last update posted 2016-09-05 (Estimated); Status verified 2016-07

CONDITIONS: Acute Respiratory Distress Syndrome (ARDS)
Keywords: Acute respiratory distress syndrome (ARDS)
MeSH Terms: conditions — Respiratory Distress Syndrome | interventions — Budesonide; Formoterol Fumarate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Budesonide and Formoterol (Experimental): Subjects randomized to this arm will receive combined standard aerosolized doses of budesonide (0.5 mg) and formoterol (20 mcg) twice daily, with at least 6 hours between doses, for 5 days for a total of 10 doses or until hospital discharge or death, with the first dose administered as soon as possible following randomization but not later than 4 hours.
  Interventions: Drug: Budesonide; Drug: Formoterol
- Placebo (Placebo Comparator): Subjects randomized to this arm will receive normal saline, the quantity, appearance and timing of the doses the same as the intervention arm.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Budesonide — Subjects will receive the standard aerosolized dose of budesonide (0.5 mg).
  Other Names: Pulmicort
  Arms: Budesonide and Formoterol
Drug: Placebo — Aerosolized normal saline will be prepared to mimic the intervention arm, with the quantity, appearance and timing of the doses the being the same.
  Arms: Placebo
Drug: Formoterol — Subjects will receive the standard aerosolized dose of formoterol (20 mcg) .
  Other Names: Foradil Aerolizer
  Arms: Budesonide and Formoterol

SUMMARY:
This study tested whether inhaled budesonide and formoterol were able to alleviate or prevent pulmonary injury when administered early in hospital course to the patients at risk for developing acute respiratory distress syndrome (ARDS). The FDA has approved many uses for budesonide and formoterol, including asthma and chronic obstructive pulmonary disease (COPD), but the use of these two drugs is experimental for ARDS.

DETAILED DESCRIPTION:
Subjects were randomized to either placebo or combined standard aerosolized doses of budesonide (0.5 mg) and formoterol (20 mcg) twice daily, with at least 6 hours between doses, for 5 calendar days for a total of 10 doses or until hospital discharge or death. Local hospital pharmacies prepared identical appearing solutions and drug was delivered by respiratory therapists blinded to randomization by using standard jet nebulizers that produce aerosol particle size within the respirable range (<5.5 microns). The first dose was administered within 4 hours after randomization.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age > 18)
* Admitted to the hospital through the emergency department (ED)
* High risk of developing ARDS (Lung Injury Prediction Score (LIPS) greater than or equal to four)

Exclusion Criteria:

* Inhaled corticosteroid and/or beta agonist treatment on admission or within 7 days prior to admission (history of asthma or COPD necessitating therapy)
* Chronic pulmonary disease requiring daytime oxygen supplementation therapy
* Systemic steroid treatment on admission or within 7 days prior to admission equivalent to more than 5 mg of prednisone daily
* Inability to obtain consent within 12 hours of hospital presentation
* Acute lung injury prior to randomization
* Receiving mechanical ventilation before current hospital admission (patient who is ventilator dependent)
* Presentation believed to be purely due to heart failure without other known risk factors for ARDS
* Allergy or other contraindication to either budesonide and/or formoterol use
* Expected hospital stay and/or survival <48 hours or admission for comfort or hospice care
* Patient, surrogate or physician not committed to full support (exception: a patient will not be excluded if he/she would receive all supportive care except for attempts at resuscitation from cardiac arrest)
* Previous enrollment in this trial.
* Co-enrollment with LIPS-A trial is not allowed.
* An active enrollment in other concomitant trial will be judged on case by case basis by PIs of both trials.
* EKG and/or clinical presentation suggestive of acute coronary ischemia
* New onset cardiac arrhythmia
* Current atrial fibrillation with ventricular rate of >110/minute
* Persistent sinus tachycardia of >130/minute despite early goal directed therapy with fluids, pressors, antibiotics and supplemental oxygen
* Pregnant patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2013-07; Primary Completion 2015-07 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emir Festic, MD, Principal Investigator — Mayo Clinic
Locations (5):
- United States (5):
  - University of Arizona, Tucson, Arizona
  - Stanford University, Stanford, California
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Beth Israel Medical Center, Boston, Massachusetts
  - Mayo Clinic in Rochester, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Festic E, Carr GE, Cartin-Ceba R, Hinds RF, Banner-Goodspeed V, Bansal V, Asuni AT, Talmor D, Rajagopalan G, Frank RD, Gajic O, Matthay MA, Levitt JE. Randomized Clinical Trial of a Combination of an Inhaled Corticosteroid and Beta Agonist in Patients at Risk of Developing the Acute Respiratory Distress Syndrome. Crit Care Med. 2017 May;45(5):798-805. doi: 10.1097/CCM.0000000000002284. PMID 28240689

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled from September 2013 to June 2015.
Period: Overall Study
Arm/Group | Budesonide and Formoterol | Placebo
Started | 30 | 31
Completed | 29 | 30
Not Completed | 1 | 1
Not completed — Screen Failure | 1 | 1

BASELINE CHARACTERISTICS:
Population: Only participants who completed the study were included in the baseline analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Budesonide and Formoterol | Placebo | Total
Number analyzed (Participants) | 29 | 30 | 59
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 71 [59 to 79] | 57 [49 to 67] | 64 [51 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 10 | 21
  Male | 18 | 20 | 38
Region of Enrollment [Number; unit: participants]
  United States | 29 | 30 | 59

OUTCOME MEASURES:

1. Primary Outcome: Change in Oxygen Saturation to Fraction of Inspired Oxygen Concentration (SpO2/FiO2) Ratio
Description: Oxygen saturation (SpO2) was measured by pulse oximetry. FiO2 is the assumed proportion of oxygen concentration participating in gas exchange in the alveoli. All S/F measurements were performed per standard operating protocol using a Venturi mask titrated to obtain an oxygen saturation of 94 ± 2% unless the patient met this goal on room air or clinical status dictated an alternative delivery mode. This outcome measure was analyzed as a longitudinal continuous variable by a mixed effect model. The formula for the calculation of SpO2/FiO2 (or S/F ratio) is %saturation/proportion of FiO2 concentration.
Time Frame: baseline to day 5 after the first treatment
Population: Intention to Treat analysis. The patient population for each day is indicated in the category by (treatment arm, placebo arm).
Measure: Median (Inter-Quartile Range); unit: SpO2/FiO2 Ratio
Arm/Group | Budesonide and Formoterol | Placebo
Number analyzed (Participants) | 29 | 30
SpO2/FiO2 Ratio
  Day 0 (29, 30) | 320 [258 to 343] | 334 [269 to 380]
  Day 1 (29, 30) | 376 [320 to 448] | 336 [269 to 448]
  Day 2 (25, 27) | 400 [343 to 457] | 332 [245 to 396]
  Day 3 (17, 24) | 396 [336 to 448] | 360 [267.5 to 450]
  Day 4 (13,19) | 448 [438 to 452] | 336 [243 to 448]
  Day 5 (6,7) | 375 [263 to 448] | 362 [248 to 452]
Statistical Analysis 1: Comparison: Budesonide and Formoterol vs Placebo; Overall p-value of the day by treatment interaction from the random effects model using a type 3 Wald test; Test type: Superiority or Other; p = 0.02, Type 3 Wald Test

2. Primary Outcome: Number of Participants Experiencing Categorical Change in Oxygen Saturation to Fraction of Inspired Oxygen Concentration (SpO2/FiO2) Ratio
Description: The data in the table below represent the greatest change from baseline observed for any one participant over all individual post-baseline measurements.
Time Frame: Days 0 - 5
Population: Intention to Treat Analysis
Measure: Number; unit: participants
Arm/Group | Budesonide and Formoterol | Placebo
Number analyzed (Participants) | 29 | 30
participants
  >20% Decrease | 0 | 8
  No change (within 20%) | 11 | 9
  > 20% Increase | 18 | 13
Statistical Analysis 1: Comparison: Budesonide and Formoterol vs Placebo; Comparison between the two arms for the 3 categories; Test type: Superiority or Other; p = 0.01, Fisher Exact

3. Secondary Outcome: Number of Subjects Who Needed Mechanical Ventilation
Time Frame: Hospital discharge, approximately day 28
Measure: Number; unit: participants
Arm/Group | Budesonide and Formoterol | Placebo
Number analyzed (Participants) | 29 | 30
participants | 6 | 16
Statistical Analysis 1: Comparison: Budesonide and Formoterol vs Placebo; Test type: Superiority or Other; p = 0.01, Chi-squared

4. Secondary Outcome: Number of Subjects Who Developed Acute Respiratory Distress Syndrome (ARDS)
Description: ARDS was defined per Berlin definition. Chest radiographs of all ventilated (non-invasive or invasive) patients were reviewed as consistent or not consistent with ARDS by the site investigator. A second adjudication was performed by an alternate principal investigator blinded to subject identification and clinical data. Final diagnosis of ARDS was determined centrally after chest radiograph adjudication was considered together with other relevant clinical data.
Time Frame: Hospital discharge, approximately day 28
Measure: Number; unit: participants
Arm/Group | Budesonide and Formoterol | Placebo
Number analyzed (Participants) | 29 | 30
participants | 0 | 7
Statistical Analysis 1: Comparison: Budesonide and Formoterol vs Placebo; Test type: Superiority or Other; p = 0.01, Fisher Exact

5. Secondary Outcome: Hospital Length of Stay
Time Frame: Baseline to Day 28
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Budesonide and Formoterol | Placebo
Number analyzed (Participants) | 29 | 30
days | 4 [3 to 7] | 8 [4 to 15]
Statistical Analysis 1: Comparison: Budesonide and Formoterol vs Placebo; Test type: Superiority or Other; p = 0.02, Cox Proportional Hazard, Fine/Gray adj

6. Secondary Outcome: Intensive Care Unit (ICU) Length of Stay
Time Frame: Baseline to Day 28
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Budesonide and Formoterol | Placebo
Number analyzed (Participants) | 29 | 30
days | 4 [1 to 17] | 6 [2 to 22]
Statistical Analysis 1: Comparison: Budesonide and Formoterol vs Placebo; Test type: Superiority or Other; p = 0.01, Kruskal-Wallis

ADVERSE EVENTS:
Time Frame: 28 days
Arm/Group | Budesonide and Formoterol | Placebo
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/30
Other Adverse Events (participants affected / at risk) | 0/29 | 1/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Budesonide and Formoterol (N=29) | Placebo (N=30)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes